CLINICAL TRIAL: NCT04660656
Title: Investigation of the Predictive Value of the Five-repetition Sit-to-stand Test (5R-STS) on the Outcome of Lumbar Back Surgery. The 5R-STS-III Study.
Brief Title: Predictive Value of the Five-repetition Sit-to-stand Test After Lumbar Spine surgerySTS-3 Study.
Acronym: 5R-STS-III
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Bergman Clinics (Other)
Responsible Party: Principal Investigator, Marc Schröder, Dr. M.L.J.F Schröder, Bergman Clinics
Other Study IDs: W20.272
Record Dates: First submitted 2020-12-01; First posted 2020-12-09 (Actual); Last update posted 2020-12-09 (Actual); Status verified 2020-12

CONDITIONS: Back Pain; Sciatica
MeSH Terms: conditions — Back Pain; Sciatica

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: 5 repetition sit-to-stand test — The sit-to-stand test with five repetitive movements is used as standard in our clinical routine to determine the patient's mobility objectively. The first measurement is performed preoperatively during surgery (baseline). The follow-up measurement is performed six weeks after the operation and one year after the operation in the clinic.
  A stool with a fixed height is used for this purpose. The patient should cross his arms over the chest and then slowly stand up until the knees are full of space. Then the patient sits down again, of course without support of the arms. The duration of the five movements is recorded using a stopwatch. The complete movement starts after the "Go" command and ends when the patient is fully upright after the fifth movement. This duration is written down as the patient's score.

SUMMARY:
Sciatica is a disabling condition that affects many people. This condition has an enormous influence on the social functioning of patients. The clinical determination of the severity of back pain is mainly done with validated questionnaires, which express the subjective pattern of complaints in a score. These usually reflect the severity of the complaints, but there is still a lack of objective and quantitative tests.

In this study, the aim is to investigate whether there is a connection between the duration of the 5R-STS test and the outcome of low back operations after one year. In other words: What is the predictive value of this test on the result of surgery?

The validated five-repetition sit-to-stand test (5R-STS) is a standardized test that has its origin in pneumology and is derived from the 1-minute sit-to-stand test. In this test, the patient stands up and sits down for 1 minute as often as possible from a chair without armrests, counting the number of movements. This not only measures how mobile the patient is, but can also say something about the condition of the heart and lungs. Recently, the 5R-STS has been described, in which the time is measured in which the patient has to stand up straight and sit down again five times from a chair.

DETAILED DESCRIPTION:
Sciatica is a disabling condition that affects many people. This condition has an enormous influence on the social functioning of patients. The clinical determination of the severity of back pain is mainly done with validated questionnaires, which express the subjective pattern of complaints in a score. These usually reflect the severity of the complaints, but there is still a lack of objective and quantitative tests.

Objective functional tests are tests in which the patient has to perform a prescribed procedure or movement while the duration of that movement is then registered. Such tests are already widely used in pneumology and cardiology, but not yet in spine surgery. So far, there are only a few objective tests for functional impairment in back pain such as the 6-minute walking test and timed-up-and-go test.

The validated five-repetition sit-to-stand test (5R-STS) is a standardized test that has its origin in pneumology and is derived from the 1-minute sit-to-stand test. In this test, the patient stands up and sits down for 1 minute as often as possible from a chair without armrests, counting the number of movements. This not only measures how mobile the patient is, but can also say something about the condition of the heart and lungs. Recently, the 5R-STS has been described, in which the time is measured in which the patient has to stand up straight and sit down again five times from a chair.

In spine disorders the 5R-STS had not yet been validated. In 2018, a research group formally validated this test for the first time in patients with lumbar hernia, lumbar canal stenosis, and degenerative spondylolisthesis.1 In this study (5R-STS-I)1 it was concluded that the 5R-STS provides additional information that the simple patient-reported outcome measures (PROMs, questionnaires) cannot demonstrate. It became clear that especially in patients with lumbar hernias two different patient groups existed, namely those with objective functional impairment (OFI) and those without OFI. This subdivision into two groups was even maintained after correction for pain levels. In a follow-up study (5R-STS-II)2 it was shown that when patients undergo the test without supervision - prior to surgery - the test results are equal.

In this study, the investigators want to assess whether there is a connection between the duration of the 5R-STS test and the outcome of low back operations after one year. In other words: What is the predictive value of this test on the result of surgery?

ELIGIBILITY:
Inclusion Criteria:

* All patients with lumbar hernias or with 1-level lumbar canal stenoses will be included (consecutive case series).

Exclusion Criteria:

* Wheelchair-bound patients, and other patients who cannot walk on their own or are bedridden, as well as pregnant patients, are excluded.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: In this study we will collect and analyze the data of 120 patients. Men and woman, all ages.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2020-11-25 (Actual); Primary Completion 2022-04-01 (Estimated); Study Completion 2022-05-01 (Estimated)

PRIMARY OUTCOMES:
5R-STS | 1 year
  The test time of the five-repetition sit-to-stand test (5R-STS) measures 12 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Marc L Schröder, MD, Principal Investigator — Bergman Clinics
Locations (2):
- Netherlands (2):
  - Department of Neurosurgery, Bergman Clinics, Naarden
  - Bergman Clinics, Naarden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: The five-repetition sit-to-stand test: evaluation of a simple and objective tool for the assessment of degenerative pathologies of the lumbar spine. — https://pubmed.ncbi.nlm.nih.gov/29957147/
- See also: Can objective functional impairment in lumbar degenerative disease be reliably assessed at home using the five-repetition sit-to-stand test? — https://pubmed.ncbi.nlm.nih.gov/30680635/